CLINICAL TRIAL: NCT07350668
Title: Comparison Between Opioid-Free Anesthesia vs Conventional Opioid-Based Anesthesia for Nasal Surgeries
Brief Title: Opioid-Free vs Opioid-Based Anesthesia for Nasal Surgeries
Acronym: Dex/Lido/Fent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Mohsen Zakaria Afia, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ms32-12-2024
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: Opioid-free anesthesia; Opioid-based anesthesia; Opioid Sparing
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: * Group OBA (Opioid-Based Anesthesia): Consisting of 30 participants, this group will receive intravenous fentanyl at a dose of 2 mcg.kg-1 three minutes prior to induction, followed by a fentanyl infusion at 0.5 mcg.kg-¹.h-¹ during the intraoperative period.
  * Group OFA (Opioid-Free Anesthesia): Comprising 30 participants, this group will receive dexmedetomidine at a dose of 1 mcg.kg-1 via intravenous infusion over 10 minutes prior to induction, followed by a continuous infusion of 0.6 mcg.kg-¹.h-¹ throughout the surgery. Intravenous lignocaine at 1.5 mg.kg-1 will be administered three minutes prior to induction, followed by an intraoperative infusion at 1.5 mg.kg-¹.h-¹.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: the study is double-blinded (patient and outcome assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dex and lido (Active Comparator): this group will receive dexmedetomidine at a dose of 1 mcg.kg-1 via intravenous infusion over 10 minutes prior to induction, followed by a continuous infusion of 0.6 mcg.kg-¹.h-¹ throughout the surgery. Intravenous lignocaine at 1.5 mg.kg-1 will be administered three minutes prior to induction, followed by an intraoperative infusion at 1.5 mg.kg-¹.h-¹.
  Interventions: Drug: dexmedetomidine and lignocaine infusion
- Fent (Active Comparator): this group will receive intravenous fentanyl at a dose of 2 mcg.kg-1 three minutes prior to induction, followed by a fentanyl infusion at 0.5 mcg.kg-¹.h-¹ during the intraoperative period.
  Interventions: Drug: Fentanyl infusion

INTERVENTIONS:
Drug: dexmedetomidine and lignocaine infusion — this group will receive dexmedetomidine at a dose of 1 mcg.kg-1 via intravenous infusion over 10 minutes prior to induction, followed by a continuous infusion of 0.6 mcg.kg-¹.h-¹ throughout the surgery. Intravenous lignocaine at 1.5 mg.kg-1 will be administered three minutes prior to induction, followed by an intraoperative infusion at 1.5 mg.kg-¹.h-¹.
  Arms: dex and lido
Drug: Fentanyl infusion — this group will receive intravenous fentanyl at a dose of 2 mcg.kg-1 three minutes prior to induction, followed by a fentanyl infusion at 0.5 mcg.kg-¹.h-¹ during the intraoperative period.
  Arms: Fent

SUMMARY:
The goal of this clinical trial is to evaluate and compare the efficacy, onset, duration of action, analgesic effect, and side effects of opioid-free anesthesia using dexmedetomidine and lignocaine versus conventional opioid-based anesthesia using fentanyl in patients undergoing nasal surgeries, including functional endoscopic sinus surgery (FESS) and septoplasty. The main questions it aims to answer are:

* What is the effect of opioid-free anesthesia vs opioid-based anesthesia on VAS score ?
* What is the effect of opioid-free anesthesia vs opioid-based anesthesia on postoperative complications including nausea and vomiting , postoperative Ramsay sedation score, amount of rescue analgesia , hemodynamic stability and patient satisfaction ? patients will be divided into two equal groups:
* Group OBA (Opioid-Based Anesthesia): Consisting of 30 participants, this group will receive intravenous fentanyl at a dose of 2 mcg.kg-1 three minutes prior to induction, followed by a fentanyl infusion at 0.5 mcg.kg-¹.h-¹ during the intraoperative period.
* Group OFA (Opioid-Free Anesthesia): Comprising 30 participants, this group will receive dexmedetomidine at a dose of 1 mcg.kg-1 via intravenous infusion over 10 minutes prior to induction, followed by a continuous infusion of 0.6 mcg.kg-¹.h-¹ throughout the surgery. Intravenous lignocaine at 1.5 mg.kg-1 will be administered three minutes prior to induction, followed by an intraoperative infusion at 1.5 mg.kg-¹.h-¹.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60, scheduled to undergo elective nasal surgeries.
* ASA (American Society of Anesthesiologists) physical status I-II.
* Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

* ASA III or above.
* Patients with a history of opioid dependence or chronic pain conditions requiring long-term opioid therapy.
* Patients with multiorgan failure, unstable hemodynamics prior to surgery, or scheduled for emergency surgery.
* Pregnant or lactating women.
* Patients with a history of severe asthma or those taking preoperative alpha-blockers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Postoperative Pain Intensity | 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 6 hours, 12 hours, and 24 hours postoperatively.
  Postoperative pain intensity will be assessed using the Visual Analog Scale for Pain (VAS), which ranges from 0 to 10, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain.
  Baseline pain score will be defined as the VAS score measured immediately after arrival to the post-anesthesia care unit (PACU). The primary outcome will be the change from baseline in VAS pain scores at each postoperative assessment time point, comparing opioid-free and opioid-based anesthesia approaches

SECONDARY OUTCOMES:
Change From Baseline in Mean Arterial Pressure | Baseline, after infusion, after induction, after intubation, 15 minutes, 30 minutes, 1 hour, immediately after extubation, 5 minutes after extubation, and 30 minutes after extubation.
  Mean arterial pressure (MAP), measured in mmHg, will be used to assess perioperative hemodynamic changes associated with opioid-free versus opioid-based anesthesia. Baseline MAP will be defined as the measurement obtained before study drug infusion. The secondary outcome will be the change from baseline in MAP at each specified time point. MAP will be calculated using the standard formula:
  MAP = (Systolic Blood Pressure + 2 × Diastolic Blood Pressure) / 3.
Change From Baseline in Heart Rate | Baseline, after infusion, after induction, after intubation, 15 minutes, 30 minutes, 1 hour, immediately after extubation, 5 minutes after extubation, and 30 minutes after extubation.
  Heart rate (HR), measured in beats per minute (bpm), will be recorded to assess perioperative hemodynamic responses. Baseline HR will be defined as the measurement obtained before study drug infusion. The secondary outcome will be the change from baseline in HR at each specified time point.
Change From Baseline in Quality of Recovery Score (QoR-40) | Preoperatively (baseline) and 24 hours postoperatively.
  Quality of recovery will be assessed using the Quality of Recovery-40 questionnaire (QoR-40), a validated patient-reported outcome measure consisting of 40 items across five domains (emotional state, physical comfort, psychological support, physical independence, and pain). The total score ranges from 40 to 200, where higher scores indicate better quality of recovery.
  Baseline QoR-40 will be defined as the score obtained preoperatively. The secondary outcome will be the change from baseline in total QoR-40 score comparing opioid-free and opioid-based anesthesia approaches.
Need for Rescue Analgesia | From the end of surgery up to 24 hours postoperatively.
  The need for rescue analgesia will be assessed during the first 24 hours postoperatively. Rescue analgesia will consist of intravenous ketorolac 30 mg, administered according to the study protocol.
  The secondary outcome will include:
  The proportion of participants requiring rescue analgesia, and
  Time to first analgesic request, defined as the time elapsed (in minutes) from the end of surgery to the first request for rescue analgesia (IV ketorolac 30 mg), and
  Total rescue analgesic consumption, defined as the total dose of ketorolac (mg) administered within the first 24 hours postoperatively.
  A higher proportion of participants requiring rescue analgesia, a shorter time to first analgesic request, and a greater total ketorolac consumption indicate worse postoperative analgesia.
Postoperative Nausea and Vomiting (PONV) | 30 minutes, 60 minutes, 90 minutes, and 2 hours postoperatively.
  The incidence and severity of postoperative nausea and vomiting (PONV) will be assessed at 30 minutes, 60 minutes, 90 minutes, and 2 hours postoperatively using a three-point scale:
  0 = none
  I = mild
  II = severe
  Both the proportion of participants experiencing PONV and the severity score at each time point will be recorded. Higher scores indicate more severe PONV.
Patient and Surgeon Satisfaction | 24 hours postoperatively.
  Patient and surgeon satisfaction with the surgical and anesthetic experience will be assessed using a five-point Likert scale, where:
  1. = Very dissatisfied
  2. = Dissatisfied
  3. = Neutral
  4. = Satisfied
  5. = Very satisfied
  Satisfaction scores will be recorded separately for patients and surgeons at 24 hours postoperatively. Higher scores indicate greater satisfaction.
Postoperative Sedation Level (Ramsay Sedation Score) | 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours postoperatively.
  Sedation levels will be assessed using the Ramsay Sedation Score (RSS), a validated scale ranging from 1 to 6, where:
  1. = Anxious and agitated or restless
  2. = Cooperative, oriented, and tranquil
  3. = Responds to commands only
  4. = Brisk response to light glabellar tap or loud auditory stimulus
  5. = Sluggish response to light glabellar tap or loud auditory stimulus
  6. = No response
  Higher scores indicate deeper sedation. Sedation will be recorded at 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours, 12 hours, and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No